CLINICAL TRIAL: NCT04285983
Title: Specified Drug Use Surveillance on Zafatek Tablets 25 mg -Surveillance on Long-Term Use of Trelagliptin Tablets in Type 2 Diabetes Mellitus Patients With Severe Renal Impairment or End-Stage Renal Failure-
Brief Title: Specified Drug-Use Survey of Trelagliptin Tablets "Survey on Long-term Use in Type 2 Diabetes Mellitus Patients With Severe Renal Impairment or End-stage Renal Disease"
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Trelagliptin-4004; jRCT1080225091 (Registry Identifier: jRCT)
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — trelagliptin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trelagliptin 25 mg: Trelagliptin 25 milligrams (mg) tablet, orally, once weekly for up to 12 months. Participants received interventions as part of routine medical care.
  Interventions: Drug: Trelagliptin

INTERVENTIONS:
Drug: Trelagliptin — Trelagliptin tablets
  Other Names: Zafatek tablets

SUMMARY:
The purpose of this study is to evaluate the long-term safety of trelagliptin tablets in patients with type 2 diabetes mellitus complicated by severe renal impairment or end-stage renal failure in the routine clinical setting.

DETAILED DESCRIPTION:
The drug being tested in this study is called trelagliptin tablet. This tablet is being tested to treat people who have type 2 diabetes mellitus complicated by severe renal impairment or end-stage renal failure.

This study is an observational (non-interventional) study and will look at the long-term safety of the trelagliptin tablet in the routine clinical setting. The planned number of observed patients will be approximately 100.

This multi-center observational trial will be conducted in Japan.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be type 2 diabetes mellitus patients meeting the following conditions: Have severe renal impairment or end-stage renal disease, with serum creatinine (mg/dL) or creatinine clearance (Ccr; mL/min) meeting the following criteria within 3 months before the start of treatment with this product

* Serum creatinine (mg/dL)*: male: > 2.4, female: > 2.0
* Ccr (mL/min): < 30 In patients with end-stage renal disease, this product may be administered irrespective of the time of hemodialysis.

  * Estimated values corresponding to the Ccr (for persons aged 60 years weighing 65 kg)

Exclusion Criteria:

1. Participants with any of the following contraindications for trelagliptin will be excluded:

1. Patient with severe ketosis, diabetic coma or pre-coma, or type 1 diabetes mellitus
2. Patient with severe infection, perioperative status, or serious trauma
3. Patient with a history of hypersensitivity to any ingredients of trelagliptin

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with type 2 diabetes mellitus complicated by severe renal impairment or end-stage renal failure as part of routine medical care.
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda Selected Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b603c4db2bf003ab4a386

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the survey at 12 investigative sites in Japan, from 1 March 2020 to 31 January 2023.
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus complicated by severe renal impairment or end-stage renal failure were enrolled. Participants received trelagliptin as part of a routine medical care.
Period: Overall Study
Arm/Group | Trelagliptin 25 mg
Started | 89
Completed | 83
Not Completed | 6
Not completed — Protocol Violation | 6

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Arm/Group | Trelagliptin 25 mg
Number analyzed (Participants) | 83
Age, Continuous [Mean (Standard Deviation); unit: Years] | 77.5 (9.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — All participants were enrolled in Japan.
  Participants
    Japan | 83
Duration of Type 2 Diabetes Mellitus [Mean (Standard Deviation); unit: Years] — Mean duration between the first diagnosis of type 2 diabetes mellitus and the start of the study was reported. Population: The number analyzed is the number of participants with data available for analysis.
  Years
    number analyzed (Participants) | 54
    (all) | 17.4 (10.08)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] — Population: The number analyzed is the number of participants with data available for analysis.
  Kilograms (kg)
    number analyzed (Participants) | 75
    (all) | 58.42 (11.611)
BMI [Mean (Standard Deviation); unit: Kilogram (kg)/meter (m)^2]] — Body Mass Index = weight (kg)/[height (m)^2] Population: The number analyzed is the number of participants with data available for analysis.
  Kilogram (kg)/meter (m)^2]
    number analyzed (Participants) | 72
    (all) | 23.04 (3.625)
Height [Mean (Standard Deviation); unit: Centimeters (cm)] — Population: The number analyzed is the number of participants with data available for analysis.
  Centimeters (cm)
    number analyzed (Participants) | 76
    (all) | 159.2 (9.88)
Healthcare Category [Count of Participants; unit: Participants] — Participants were categorized as outpatient and inpatient.
  Participants
    Outpatient | 83
    Inpatient | 0
Dialysis Treatment Status [Count of Participants; unit: Participants]
  Had No Dialysis Treatment | 63
  Had Dialysis Treatment | 20
Predisposition to Hypersensitivity [Count of Participants; unit: Participants] — Number of participants who had or did not have a liability or tendency to suffer from hypersensitivity was reported. Unknown: Data could not be collected.
  Participants
    Had No Predisposition to Hypersensitivity | 63
    Had Predisposition to Hypersensitivity | 18
    Unknown | 2
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had No Medical Complications | 0
    Had Medical Complications | 83
Medical History [Count of Participants; unit: Participants] — Medical history defined as a disease or a health condition for each participant before start of the study. Medical history was classified as congenital anomalies, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, GI disorders, hepatic and biliary disorders, renal disease and other medical history. Other medical history included all medical history except for those mentioned above. Unknown: Data could not be collected.
  Participants
    Had No Medical History | 18
    Had Medical History | 60
    Unknown | 5
Smoking Classification [Count of Participants; unit: Participants] — Unknown: Data could not be collected.
  Participants
    Never Smoked | 43
    Current Smoker | 10
    Ex-Smoker | 22
    Unknown | 8
Alcohol Classification [Count of Participants; unit: Participants] — Participants who answered Yes or No for a question "Drink Alcohol Almost Every Day?" were reported. Unknown: Data could not be collected.
  Participants
    No | 16
    Yes | 60
    Unknown | 7
Hepatic Impairment [Count of Participants; unit: Participants]
  Had No Hepatic Impairment | 69
  Had Hepatic Impairment | 14
Glycated hemoglobin A1c (HbA1c) [National Glycohemoglobin Standardization Program (NGSP)] [Mean (Standard Deviation); unit: Percent] — Population: The number analyzed is the number of participants with data available for analysis.
  Percent
    number analyzed (Participants) | 67
    (all) | 6.71 (0.956)
Fasting Blood Glucose [Mean (Standard Deviation); unit: milligram (mg)/deciliter (dL)] — Population: The number analyzed is the number of participants with data available for analysis.
  milligram (mg)/deciliter (dL)
    number analyzed (Participants) | 31
    (all) | 124.5 (40.48)
Serum Creatinine Value Within 3 Months Before Start of Treatment with the Study Drug [Mean (Standard Deviation); unit: mg/dL] — Population: The number analyzed is the number of participants with data available for analysis.
  mg/dL
    number analyzed (Participants) | 57
    (all) | 2.399 (1.1757)
Creatinine Clearance Within 3 Months Before Start of Treatment with the Study Drug [Mean (Standard Deviation); unit: milliliter (mL)/minute (min)] — Population: The number analyzed is the number of participants with data available for analysis.
  milliliter (mL)/minute (min)
    number analyzed (Participants) | 47
    (all) | 22.915 (5.2967)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had One or More Adverse Drug Reactions (ADRs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. Adverse drug reaction refers to AE related to administered drug.
Time Frame: Up to Month 12
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Trelagliptin 25 mg
Number analyzed (Participants) | 83
Participants | 6

2. Primary Outcome: Number of Participants Who Had One or More Serious ADRs
Description: AE is defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug. A serious adverse event is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above mentioned criteria. Among these, events which are considered possibly associated with a medicinal product are defined as adverse drug reactions.
Time Frame: Up to Month 12
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Trelagliptin 25 mg
Number analyzed (Participants) | 83
Participants | 2

3. Primary Outcome: Number of Participants Who Had One or More Hypoglycemia of Serious ADRs and the Other ADRs
Description: Number of participants who had one or more hypoglycemia of serious ADRs and the other ADRs (non-serious ADRs) were reported. AE is defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug. A serious adverse event is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above mentioned criteria. Among these, events which are considered possibly associated with a medicinal product are defined as adverse drug reactions.
Time Frame: Up to Month 12
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Trelagliptin 25 mg
Number analyzed (Participants) | 83
Participants
  Serious ADRs | 0
  Other ADRs | 1

4. Primary Outcome: Number of Participants Who Had One or More Infection of Serious ADRs and the Other ADRs
Description: Number of participants who had one or more infection of serious ADRs and the other ADRs (non-serious ADRs) were reported. AE is defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug. A serious adverse event is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above mentioned criteria. Among these, events which are considered possibly associated with a medicinal product are defined as adverse drug reactions.
Time Frame: Up to Month 12
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Trelagliptin 25 mg
Number analyzed (Participants) | 83
Participants
  Serious ADRs | 0
  Other ADRs | 0

ADVERSE EVENTS:
Time Frame: Up to Month 12
Description: At each visit the investigator had to document any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to the survey treatment.
Arm/Group | Trelagliptin 25 mg
All-Cause Mortality (participants affected / at risk) | 5/83
Serious Adverse Events (participants affected / at risk) | 33/83
Other Adverse Events (participants affected / at risk) | 10/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trelagliptin 25 mg (N=83)
Herpes zoster (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Device related infection (Infections and infestations) | 1
Nephrogenic anaemia (Blood and lymphatic system disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Ketoacidosis (Metabolism and nutrition disorders) | 1
Carotid artery stenosis (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Cholinergic syndrome (Nervous system disorders) | 1
Cataract (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Vitreous haemorrhage (Eye disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 2
Angina pectoris (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 2
Cardiac failure chronic (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Erosive oesophagitis (Gastrointestinal disorders) | 1
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Neurogenic bladder (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 3
Chronic kidney disease (Renal and urinary disorders) | 1
Death (General disorders) | 2 — The reasons of events are not determined because assessment findings were insufficient to specify the reason.
Fall (Injury, poisoning and procedural complications) | 3
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Shunt occlusion (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Shunt stenosis (Injury, poisoning and procedural complications) | 4
Device pacing issue (Product Issues) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trelagliptin 25 mg (N=83)
Periodontitis (Infections and infestations) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Hypertension (Vascular disorders) | 4
Hepatic function abnorma (Hepatobiliary disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/83/NCT04285983/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-26): https://cdn.clinicaltrials.gov/large-docs/83/NCT04285983/SAP_001.pdf